CLINICAL TRIAL: NCT01826981
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Efficacy and Safety of Sofosbuvir Containing Regimens for the Treatment of Chronic HCV Infection
Brief Title: Efficacy and Safety of Sofosbuvir Containing Regimens for the Treatment of Chronic HCV Infection in Participants With Chronic Genotype 1, 2, 3, or 6 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0122
Record Dates: First submitted 2013-04-01; First posted 2013-04-09 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir; peginterferon alfa-2a; GS-9669; velpatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- Cohort 1,Group 1: LDV/SOF + RBV 12 wk (GT1 SOF retreatment) (Experimental): LDV/SOF + RBV for 12 weeks in participants with genotype 1 HCV infection and who failed to achieve sustained virologic response (SVR) in a previous Gilead sofosbuvir study
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort 1,Group 2:SOF+Peg-IFN+RBV 12 wk (GT2,3 SOF retreatment) (Experimental): SOF + PEG + RBV for 12 weeks in participants with genotype 2 or 3 HCV infection and who failed to achieve SVR in a previous Gilead sofosbuvir study
  Interventions: Drug: SOF; Drug: RBV; Drug: Peg-IFN
- Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, liver disease) (Experimental): LDV/SOF+RBV for 12 weeks in treatment-experienced participants with genotype 1 HCV infection and advanced liver fibrosis or compensated liver fibrosis
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort 2,Group 2: LDV/SOF+GS-9669 12wk (GT1 TE, liver disease) (Experimental): LDV/SOF + GS-9669 for 12 weeks in treatment-experienced participants with genotype 1 HCV infection and advanced liver fibrosis or compensated liver fibrosis
  Interventions: Drug: LDV/SOF; Drug: GS-9669
- Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) (Experimental): LDV/SOF for 12 weeks in treatment-naive participants with genotype 3 HCV infection
  Interventions: Drug: LDV/SOF
- Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) (Experimental): LDV/SOF + RBV for 12 weeks in treatment-naive participants with genotype 3 HCV infection
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) (Experimental): LDV/SOF for 12 weeks in treatment-naive or treatment-experienced participants with genotype 6 HCV infection
  Interventions: Drug: LDV/SOF
- Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) (Experimental): LDV/SOF + RBV for 12 weeks in treatment-experienced participants with genotype 3 HCV infection
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort 3,Group 1: LDV/SOF 12 wk (GT1 cirrhotic CPT B) (Experimental): LDV/SOF for 12 weeks in participants with genotype 1 HCV infection and Child-Pugh Turcotte (CPT) B cirrhosis
  Interventions: Drug: LDV/SOF
- Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN noncirrhotic) (Experimental): SOF+VEL (25 mg) for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
  Interventions: Drug: SOF; Drug: VEL
- Cohort 4,Group 2:SOF+VEL 25mg+RBV 8 wk (GT3 TN noncirrhotic) (Experimental): SOF+VEL(25 mg)+RBV for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
  Interventions: Drug: SOF; Drug: RBV; Drug: VEL
- Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN noncirrhotic) (Experimental): SOF+VEL (100 mg) for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
  Interventions: Drug: SOF; Drug: VEL
- Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN noncirrhotic) (Experimental): SOF+VEL (100 mg)+RBV for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
  Interventions: Drug: SOF; Drug: RBV; Drug: VEL
- Cohort 5,Group 1: LDV/SOF + RBV 24 wk (SOF retreatment) (Experimental): LDV/SOF+RBV for 24 weeks in participants with genotype 1, 2, 3, or 6 HCV infection and who failed to achieve SVR in a previous Gilead sofosbuvir study
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HBV coinfection) (Experimental): LDV/SOF for 12 weeks in participants with genotype 1 HCV and hepatitis B virus (HBV) coinfection
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — Ledipasvir/sofosbuvir (LDV/SOF) (90 /400 mg) fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
  Arms: Cohort 1,Group 1: LDV/SOF + RBV 12 wk (GT1 SOF retreatment); Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, liver disease); Cohort 2,Group 2: LDV/SOF+GS-9669 12wk (GT1 TE, liver disease); Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN); Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN); Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN); Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE); Cohort 3,Group 1: LDV/SOF 12 wk (GT1 cirrhotic CPT B); Cohort 5,Group 1: LDV/SOF + RBV 24 wk (SOF retreatment); Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HBV coinfection)
Drug: SOF — SOF 400 mg tablet administered orally once daily
  Other Names: GS-7977; Sovaldi®
  Arms: Cohort 1,Group 2:SOF+Peg-IFN+RBV 12 wk (GT2,3 SOF retreatment); Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 2:SOF+VEL 25mg+RBV 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN noncirrhotic)
Drug: RBV — Ribavirin (RBV) 200 mg tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: Cohort 1,Group 1: LDV/SOF + RBV 12 wk (GT1 SOF retreatment); Cohort 1,Group 2:SOF+Peg-IFN+RBV 12 wk (GT2,3 SOF retreatment); Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, liver disease); Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN); Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE); Cohort 4,Group 2:SOF+VEL 25mg+RBV 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN noncirrhotic); Cohort 5,Group 1: LDV/SOF + RBV 24 wk (SOF retreatment)
Drug: Peg-IFN — pegylated interferon (Peg-IFN) 180 µg administered subcutaneously once weekly
  Other Names: Pegasys®
  Arms: Cohort 1,Group 2:SOF+Peg-IFN+RBV 12 wk (GT2,3 SOF retreatment)
Drug: GS-9669 — GS-9669 500 mg (2 × 250 mg tablet) administered orally once daily
  Arms: Cohort 2,Group 2: LDV/SOF+GS-9669 12wk (GT1 TE, liver disease)
Drug: VEL — Velpatasvir (VEL) tablet(s) administered orally once daily
  Other Names: GS-5816
  Arms: Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 2:SOF+VEL 25mg+RBV 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN noncirrhotic); Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN noncirrhotic)

SUMMARY:
The purpose of this study is to evaluate the antiviral efficacy, safety, tolerability of combination therapy with sofosbuvir (SOF) containing regimens for the treatment of chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1, 2, 3, or 6 HCV infection
* Cirrhosis determination; a liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hyland, DPhil, Study Director — Gilead Sciences
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies Ltd., Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Gane EJ, Hyland RH, An D, Svarovskaia E, Pang PS, Brainard D, Stedman CA. Efficacy of ledipasvir and sofosbuvir, with or without ribavirin, for 12 weeks in patients with HCV genotype 3 or 6 infection. Gastroenterology. 2015 Nov;149(6):1454-1461.e1. doi: 10.1053/j.gastro.2015.07.063. Epub 2015 Aug 7. PMID 26261007
- [Result] Gane EJ, Hyland RH, An D, Svarovskaia ES, Brainard D, McHutchison JG. Ledipasvir and sofosbuvir for HCV infection in patients coinfected with HBV. Antivir Ther. 2016;21(7):605-609. doi: 10.3851/IMP3066. Epub 2016 Jul 1. PMID 27367295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 2 study sites in New Zealand. The first participant was screened on 3 April 2016. The last study visit occurred on 25 May 2015.
Pre-assignment Details: 446 participants were screened.
Groups:
- Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment): Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 12 weeks in participants with genotype 1 HCV infection and who failed to achieve SVR in a previous Gilead sofosbuvir study.
- Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment): SOF 400 mg once daily+ pegylated interferon (PEG-IFN) 180 µg once weekly+weight-based RBV (1000-1200 mg in a divided daily dose) for 12 weeks in participants with genotype 2 or 3 HCV infection and who failed to achieve SVR in a previous Gilead sofosbuvir study
- Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease): LDV/SOF (90/400 mg) once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 12 weeks in treatment-experienced (TE) participants with genotype 1 HCV infection and advanced liver fibrosis or compensated liver fibrosis
- Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease: LDV/SOF (90/400 mg) once daily + GS-9669 500 mg once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection and advanced liver fibrosis or compensated liver fibrosis
- Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN): LDV/SOF (90/400 mg) once daily for 12 weeks in treatment-naive (TN) participants with genotype 3 HCV infection
- Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN): LDV/SOF (90/400 mg) once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 12 weeks in treatment-naive participants with genotype 3 HCV infection
- Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN): LDV/SOF (90/400 mg) once daily for 12 weeks in treatment-naive or treatment-experienced participants with genotype 6 HCV infection
- Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE): LDV/SOF (90/400 mg) once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 12 weeks in treatment-experienced participants with genotype 3 HCV infection
- Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B): LDV/SOF (90/400 mg) once daily for 12 weeks in participants with genotype 1 HCV infection and Child Pugh-Turcotte (CPT) B cirrhosis
- Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic): Sofosbuvir (SOF) 400 mg once daily+Velpatasvir (VEL) 25 mg once daily for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
- Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic): SOF 400 mg once daily +VEL 25 mg once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
- Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic): SOF 400 mg once daily+VEL 100 mg once daily for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
- Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic): SOF 400 mg once daily+VEL 100 mg once daily + weight-based RBV (1000-1200 mg in a divided daily dose) for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
- Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment): LDV/SOF (90/400 mg) once daily+weight-based RBV (1000-1200 mg in a divided daily dose) for 24 weeks in participants with genotype 1 or 3 HCV infection and who failed to achieve SVR in a previous Gilead sofosbuvir study
- Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection): LDV/SOF (90/400 mg) once daily for 12 weeks in participants with genotype 1 HCV and hepatitis B virus (HBV) coinfection
Period: Overall Study
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Started | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 51 | 20 | 27 | 24 | 27 | 26 | 20 | 8
Completed | 19 | 9 | 25 | 26 | 18 | 25 | 24 | 40 | 13 | 26 | 22 | 25 | 25 | 15 | 8
Not Completed | 0 | 1 | 0 | 0 | 7 | 1 | 1 | 11 | 7 | 1 | 2 | 2 | 1 | 5 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 8 | 7 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Upper G-I Haemorrhage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Enrolled/Randomized but Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Participants who were randomized and received at least 1 dose of study drug.
Groups:
- Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B): LDV/SOF (90/400 mg) once daily for 12 weeks in participants with genotype 1 HCV infection and CPT B cirrhosis
- Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic): SOF 400 mg once daily+VEL 25 mg once daily for 8 weeks in treatment-naive noncirrhotic participants with genotype 3 HCV infection
- Total: Total of all reporting groups
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection) | Total
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 27 | 26 | 20 | 8 | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (6.1) | 49 (12.5) | 56 (5.3) | 55 (6.7) | 43 (10.2) | 48 (9.2) | 51 (13.9) | 52 (8.2) | 56 (5.5) | 48 (7.9) | 47 (7.9) | 50 (10.2) | 47 (10.3) | 54 (7.0) | 53 (6.9) | 50.7 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 10 | 11 | 12 | 15 | 9 | 11 | 3 | 10 | 6 | 10 | 15 | 2 | 2 | 124
  Male | 13 | 8 | 15 | 15 | 13 | 11 | 16 | 39 | 17 | 17 | 18 | 17 | 11 | 18 | 6 | 234
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 9 | 22 | 24 | 22 | 23 | 3 | 40 | 17 | 20 | 20 | 20 | 19 | 18 | 3 | 278
  Asian | 0 | 0 | 1 | 0 | 1 | 1 | 22 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 5 | 2 | 5 | 2 | 3 | 6 | 1 | 4 | 34
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 27 | 26 | 20 | 8 | 358
HCV Genotype [Number; unit: participants]
  1b with possible mixed infection with Genotype 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Genotype 1a | 16 | 0 | 15 | 22 | 0 | 0 | 0 | 0 | 18 | 0 | 0 | 0 | 0 | 9 | 6 | 86
  Genotype 1a with possible 6 (subtypes c - l) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Genotype 1b | 2 | 0 | 9 | 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 19
  Genotype 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 7
  Genotype 3a | 0 | 10 | 0 | 0 | 24 | 25 | 0 | 46 | 0 | 25 | 22 | 27 | 26 | 10 | 0 | 215
  Genotype 3k | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Genotype 6 (subtypes c - l) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17
  Genotype 6a or 6b | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Indeterminate genotype. Sequencing indicates GT3a | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Indeterminate pattern. Sequencing indicates GT3k | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cirrhosis Status [Number; unit: participants]
  No | 18 | 9 | 7 | 9 | 21 | 20 | 23 | 28 | 0 | 27 | 24 | 27 | 26 | 6 | 6 | 251
  Yes | 1 | 1 | 18 | 17 | 4 | 6 | 2 | 22 | 20 | 0 | 0 | 0 | 0 | 14 | 2 | 107
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 3 | 6 | 4 | 9 | 15 | 20 | 18 | 7 | 10 | 6 | 15 | 14 | 7 | 7 | 145
    CT | 12 | 5 | 12 | 19 | 10 | 6 | 5 | 27 | 6 | 13 | 15 | 11 | 10 | 7 | 1 | 159
    TT | 3 | 2 | 7 | 3 | 6 | 5 | 0 | 5 | 7 | 4 | 3 | 1 | 2 | 6 | 0 | 54
HCV RNA [Median (Standard Deviation); unit: log 10 IU/mL] | 6.3 (0.51) | 6.5 (0.63) | 6.5 (0.39) | 6.1 (0.69) | 6.3 (0.88) | 6.3 (0.87) | 6.7 (0.67) | 6.3 (0.76) | 6.0 (0.48) | 5.9 (0.86) | 6.3 (0.69) | 6.0 (0.71) | 6.2 (0.92) | 6.0 (0.48) | 6.0 (10.9) | 6.2 (0.76)
HCV RNA Category [Number; unit: IU/mL]
  < 800,000 | 3 | 1 | 2 | 9 | 9 | 6 | 2 | 15 | 5 | 14 | 10 | 11 | 7 | 6 | 2 | 102
  >= 800,000 | 16 | 9 | 23 | 17 | 16 | 20 | 23 | 35 | 15 | 13 | 14 | 16 | 19 | 14 | 6 | 256

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full analysis set: Participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 27 | 26 | 20 | 8
percentage of participants | 100 | 90 | 100 | 100 | 64.0 | 100 | 96.0 | 82.0 | 65.0 | 100 | 87.5 | 96.3 | 100.0 | 75 | 100

2. Primary Outcome: Percentage of Participants With Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 27 | 26 | 20 | 8
Percentage of participants | 0 | 0 | 4.0 | 0 | 4.0 | 0 | 0 | 2.0 | 0 | 0 | 4.2 | 0 | 3.8 | 5.0 | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) While on Treatment
Time Frame: Weeks 1 and 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 26 | 26 | 20 | 8
percentage of participants
  Week 1 | 15.8 | 30.0 | 4.0 | 11.5 | 20.0 | 11.5 | 12.0 | 12.0 | 0 | 33.3 | 4.2 | 26.9 | 19.2 | 15.0 | 12.5
  Week 2 | 63.2 | 50.0 | 44.0 | 53.8 | 64.0 | 61.5 | 56.0 | 52.0 | 25.0 | 70.4 | 66.7 | 65.4 | 69.2 | 45.0 | 75.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) While on Treatment
Time Frame: Weeks 4, 6, and 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 24 | 26 | 25 | 50 | 20 | 27 | 23 | 26 | 26 | 20 | 8
percentage of participants
  Week 4 | 100.0 | 100.0 | 84.0 | 92.3 | 95.8 | 88.5 | 96.0 | 96.0 | 75.0 | 96.3 | 95.7 | 92.3 | 96.2 | 75.0 | 87.5
  Week 6 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 96.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 90.0 | 100.0
  Week 8 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 90.0 | 100.0

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) While on Treatment
Time Frame: Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 23 | 25 | 24 | 50 | 20 | 20 | 8
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 98.0 | 100.0 | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) While on Treatment
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 23 | 24 | 24 | 50 | 20 | 20 | 8
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 98.0 | 100.0 | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) While on Treatment
Time Frame: Weeks 16, 20, and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment)
Number analyzed (Participants) | 20
percentage of participants
  Week 16 | 100.0
  Week 20 | 100.0
  Week 24 | 100.0

8. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) at 2, 4, 8, and 24 Weeks After Discontinuation of Therapy (SVR2, SVR4, SVR8, and SVR 24)
Time Frame: Posttreatment Weeks 2, 4, 8, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 24 | 26 | 25 | 50 | 20 | 27 | 23 | 26 | 26 | 20 | 8
percentage of participants
  SVR2 | 100.0 | 100.0 | 100.0 | 100.0 | 72.0 | 100.0 | 100.0 | 90.0 | 95.0 | 100.0 | 87.5 | 96.3 | 100.0 | 95.0 | 100.0
  SVR4 | 100.0 | 100.0 | 84.0 | 92.3 | 95.8 | 88.5 | 96.0 | 96.0 | 75.0 | 96.3 | 95.7 | 92.3 | 96.2 | 75.0 | 87.5
  SVR8 | 100.0 | 90.0 | 100.0 | 100.0 | 64.0 | 100.0 | 96.0 | 82.0 | 65.0 | 100.0 | 87.5 | 96.3 | 100.0 | 80.0 | 100.0
  SVR24 | 100.0 | 90.0 | 100.0 | 100.0 | 64.0 | 100.0 | 96.0 | 82.0 | 65.0 | 100.0 | 87.5 | 96.3 | 100.0 | 75.0 | 100.0

9. Secondary Outcome: For Cohort 6, Percentage of Participants With HCV RNA < LLOQ (15 IU/mL) at 16 and 20 Weeks After Discontinuation of Therapy (SVR16 and SVR 20)
Time Frame: Posttreatment Weeks 16 and 20
Population: Full Analysis Set included the participants who were randomized into Cohort 6 and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 8
percentage of participants
  SVR16 | 100
  SVR20 | 100

10. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 25 | 26 | 25 | 50 | 20 | 27 | 24 | 27 | 26 | 20 | 8
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse is defined as HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection)
Number analyzed (Participants) | 19 | 10 | 25 | 26 | 24 | 26 | 25 | 50 | 20 | 27 | 23 | 26 | 26 | 20 | 8
percentage of participants | 0 | 10.0 | 0 | 0 | 33.3 | 0 | 4.0 | 16.3 | 35.0 | 0 | 8.7 | 0 | 0 | 15.0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/10 | 1/25 | 0/26 | 4/25 | 0/26 | 1/25 | 1/50 | 2/20 | 3/20 | 0/8 | 1/27 | 0/24 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 17/19 | 10/10 | 24/25 | 24/26 | 24/25 | 23/26 | 21/25 | 43/50 | 19/20 | 17/20 | 6/8 | 18/27 | 18/24 | 22/27 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) (N=19) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) (N=10) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) (N=25) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease (N=26) | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) (N=25) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) (N=26) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) (N=25) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) (N=50) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) (N=20) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) (N=20) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection) (N=8) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) (N=27) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) (N=24) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) (N=27) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) (N=26)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Choroidal effusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lens dislocation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1,Group 1: LDV/SOF+RBV 12 wk (GT1 SOF Retreatment) (N=19) | Cohort 1,Group 2: SOF+Peg+RBV 12 wk (GT2,3 SOF Retreatment) (N=10) | Cohort 2,Group 1: LDV/SOF+RBV 12 wk (GT 1 TE, Liver Disease) (N=25) | Cohort 2,Group 2: LDV/SOF+GS-9669 12 wk (GT1 TE, Liver Disease (N=26) | Cohort 2,Group 3: LDV/SOF 12 wk (GT3 TN) (N=25) | Cohort 2,Group 4: LDV/SOF+RBV 12 wk (GT3 TN) (N=26) | Cohort 2,Group 5: LDV/SOF 12 wk (GT6 TE/TN) (N=25) | Cohort 2,Group 6: LDV/SOF+RBV 12 wk (GT3 TE) (N=50) | Cohort 3,Group 1: LDV/SOF 12 wk (GT1 Cirrhotic CPT B) (N=20) | Cohort 5,Group 1: LDV/SOF+RBV 24 wk (GT1/3 SOF Retreatment) (N=20) | Cohort 6,Group 1: LDV/SOF 12 wk (GT1, HCV and HBV Coinfection) (N=8) | Cohort 4,Group 1: SOF+VEL 25mg 8 wk (GT3 TN Noncirrhotic) (N=27) | Cohort 4,Group 2: SOF+VEL 25mg+RBV 8 wk (GT3 TN Noncirrhotic) (N=24) | Cohort 4,Group 3: SOF+VEL 100mg 8 wk (GT3 TN Noncirrhotic) (N=27) | Cohort 4,Group 4: SOF+VEL 100mg+RBV 8 wk (GT3 TN Noncirrhotic) (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid thickening (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 3 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 2 | 0 | 4 | 4 | 0 | 2 | 0 | 2 | 2 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 7 | 11 | 9 | 4 | 0 | 5 | 3 | 1 | 0 | 4 | 1 | 4 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 3 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 4 | 2 | 0
Catheter site bruise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 5 | 9 | 5 | 2 | 6 | 13 | 4 | 4 | 2 | 5 | 3 | 4 | 7
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 0 | 6 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 8 | 5 | 9 | 9 | 6 | 9 | 8 | 6 | 2 | 1 | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 5 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chest crushing (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 4 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 2 | 10 | 9 | 10 | 8 | 2 | 13 | 4 | 3 | 0 | 6 | 5 | 3 | 4
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 1 | 3 | 3
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 7 | 2 | 7 | 1 | 3 | 3 | 0 | 10 | 3 | 1 | 0 | 0 | 3 | 6 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 0 | 3 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2 | 1 | 1 | 2 | 7 | 1 | 3 | 0 | 0 | 3 | 2 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years